CLINICAL TRIAL: NCT00017862
Title: A Pilot Phase II Study of the Efficacy of Humanized Anti-IL5 Antibody (SCH55700) in Reducing Eosinophilia in Patients With Hypereosinophilic Syndrome or Eosinophilic Gastroenteritis Refractory to or Intolerant of Conventional Therapy
Brief Title: Anti-Interleukin-5 Antibody to Treat Hypereosinophilic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010155; 01-I-0155
Record Dates: First submitted 2001-06-15; First posted 2002-04-29 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-06

CONDITIONS: Hypereosinophilic Syndrome
Keywords: Eosinophils; Monoclonal Antibody; Hypereosinophilia; Biologicals; Hypereosinophilic Syndrome
MeSH Terms: conditions — Hypereosinophilic Syndrome; Eosinophilia | interventions — reslizumab

INTERVENTIONS:
Drug: SCH55700

SUMMARY:
This study will examine the safety and effectiveness of a single dose of anti-interleukin-5 antibody (SCH 55700) in reducing the number of eosinophils (a type of white blood cell) in patients with hypereosinophilic syndrome. Patients with this disease have too many eosinophils in the blood and in body tissues, which cause damage to the affected organs-most commonly the heart, nerves and skin. SCH 55700 is an antibody to interleukin 5-a hormone-like substance produced by white blood cells that plays a significant role in eosinophilia. SCH 55700 has lowered eosinophilia blood counts in patients with asthma and reduced the number of these cells in tissues of animals with asthma.

Patients with hypereosinophilic syndrome 18 years of age and older who have not responded to standard therapy with steroids, interferon and hydroxyurea or cannot take these drugs may be eligible for this study. Candidates will be screened with a medical history, physical examination, eye examination, and blood tests. Depending on the patient's symptoms, other diagnostic tests may be done, including studies of the eyes, lungs, skin, nerves or heart. Skin biopsy and bronchoalveolar lavage may be included in the diagnostic evaluation. For the skin biopsy, a small area about 1/3 inch in diameter is numbed and a small core of skin is surgically removed for study under the microscope. Bronchoalveolar lavage involves inserting a catheter (flexible tube) into the lungs to instill saline (salt water) and obtain a tissue sample. This test will be done only if clinically necessary.

Those enrolled in the study will be admitted to the NIH Clinical Center for a single dose of SCH 55700, injected into an arm vein. They will be monitored in the hospital for at least 72 hours for changes in eosinophil count and side effects of the injection. After discharge, laboratory tests will be done weekly for the first month, either at the Clinical Center or by the patient's local physician. Follow-up visits will then be scheduled monthly for 1 year or until the patient's eosinophil count returns to pre-treatment levels for 2 consecutive months. Follow-up visits will include a history, physical examination and blood tests, including studies on how immune cells and other substances in the blood activate or stimulate eosinophilia. A chest X-ray, electrocardiogram and pulmonary function tests will be done at 1, 3, 6 and 12 months to evaluate organ damage. Other tests may be done if medically indicated.

Bone marrow biopsy and aspiration will be done before receiving SCH 55700 and one month after the injection to evaluate the effects of SCH 55700 on eosinophil production in the bone marrow. For this test, an area of skin and bone is numbed and a very sharp needle is used to withdraw a sample of the bone marrow. Leukapheresis will also be done before and 1 month after SCH 55700 treatment to obtain cells for studying the effect of SCH 55700 on eosinophil activation, function and survival. For this procedure, whole blood is collected through a needle in an arm vein. The blood circulates through a machine that separates it into its components. The white cells are then removed, and the rest of the blood is returned to the body, either through the same needle used to draw the blood or through a second needle placed in the other arm.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of humanized monoclonal anti-IL5 antibody, SCH 55700 in reducing peripheral blood eosinophilia in patients with either hypereosinophilic syndrome or eosinophilic gastroenteritis. Patients with hypereosinophilic syndrome refractory to or intolerant of therapy with conventional therapy (steroids, hydroxyurea and interferon alpha) will be admitted on this protocol. Additionally, subjects with eosinophilic gastroenteritis refractory or intolerant to conventional therapy (systemic glucocorticoids) will be admitted on this protocol. A thorough clinical evaluation will be performed with emphasis on potential sequelae of eosinophil-mediated tissue damage. A baseline bone marrow will be obtained to exclude neoplasia and to assess the degree and nature of eosinophilipoiesis. Blood cells and/or serum will also be collected to provide reagents (such as DNA, RNA, and specific antibodies) for use in the laboratory to address issues related to the immunologic basis of FHES and GE as well as their pathogenesis and treatment. Following intravenous administration of a single 1 mg/kg dose of the humanized monoclonal anti-IL5 antibody, SCH 55700, patients will be followed in an inpatient setting for a minimum of 72 hours for monitoring of adverse effects secondary to the infusion. Followup visits will be scheduled monthly for 1 year or until the peripheral eosinophil count returns to baseline. Patients showing a reduction in eosinophilia and evidence of clinical improvement will be eligible to receive 5 additional doses of 1 mg/kg of SCH 55700 at monthly intervals.

ELIGIBILITY:
INCLUSION CRITERIA - HES:

All subjects must meet the established diagnostic criteria for idiopathic hypereosinophilic syndrome: eosinophilia greater than 1,500/mm3 on two occasions at least 6 months apart, no known etiology for the eosinophilia despite careful clinical evaluation, evidence of end organ damage (histologic evidence of tissue infiltration by eosinophils and/or objective evidence of clinical pathology in any organ system that is temporarily associated with eosinophilia and not clearly attributable to another cause).

All subjects must be at least 18 years of age.

Failure of or contraindication to treatment with steroids, interferon alpha and hydroxyurea

Negative serum beta-hCG within 24 hours of drug administration for women of childbearing potential must to exclude early pregnancy

Agree to practice abstinence or effective contraception for 6 months following administration of the study drug

INCLUSION CRITERIA - EG:

All subjects must meet the established diagnostic criteria for eosinophilic gastroenteritis: gastrointestinal symptoms, histologic evidence of gastrointestinal tissue infiltration by eosinophils with greater than or equal to 25 eosinophils per high powered field, no known etiology for the eosinophilia despite careful clinical evaluation

Eosinophilia greater than 860/mm3 on two occasions at least 6 months apart

Evidence of hypersensitivity to foods or aeroallergens as determined by skin or RAST testing

All subjects must be at least 18 years of age.

Failure of or contraindication to treatment with steroids.

Negative serum beta-hCG within 24 hours of drug administration for women of childbearing potential must to exclude early pregnancy

Agree to practice abstinence or effective contraception for 6 months following administration of the study drug

EXCLUSION CRITERIA - HES and GE:

Pregnant or nursing women

HIV positivity or other known immunodeficiency

Use of any other investigational agent within 30 days of the study

Any condition that, in the investigator's opinion, places the patient at undue risk by participating in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2001-06; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Aractingi S, Janin A, Zini JM, Gauthier MS, Chauvenet L, Tobelem G, Prin L, Chosidow O, Frances C. Specific mucosal erosions in hypereosinophilic syndrome. Evidence for eosinophil protein deposition. Arch Dermatol. 1996 May;132(5):535-41. PMID 8624150
- [Background] Fauci AS, Harley JB, Roberts WC, Ferrans VJ, Gralnick HR, Bjornson BH. NIH conference. The idiopathic hypereosinophilic syndrome. Clinical, pathophysiologic, and therapeutic considerations. Ann Intern Med. 1982 Jul;97(1):78-92. doi: 10.7326/0003-4819-97-1-78. PMID 7046556
- [Background] Weller PF, Bubley GJ. The idiopathic hypereosinophilic syndrome. Blood. 1994 May 15;83(10):2759-79. No abstract available. PMID 8180373